CLINICAL TRIAL: NCT03794323
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses of BI 764122 (Single-blind, Partially Randomised, Placebo-controlled, Parallel (Sequential) Group Design) and the Effect of Food on BI 764122 (Open-label, Randomised, Single-dose, Two-period, Two-sequence Crossover Design) in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Find Out How Well Different Doses of BI 764122 Are Tolerated and Whether Food Affects the Amount of BI 764122 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1430-0001; 2018-003604-39 (EudraCT Number)
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- SRD part: BI 764122 4 mg (Experimental): 4 uncoated tablets of 1 milligram (mg) BI 764122 (total: 4 mg) were administered as single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h). Single rising dose (SRD) part.
  Interventions: Drug: BI 764122
- SRD part: BI 764122 12 mg (Experimental): 1 film-coated tablet of 10 mg and 2 uncoated tablets of 1 mg BI 764122 (total: 12 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
  Interventions: Drug: BI 764122
- SRD part: BI 764122 25 mg (Experimental): 2 film-coated tablets of 10 mg and 5 uncoated tablets of 1 mg BI 764122 (total: 25 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
  Interventions: Drug: BI 764122
- SRD part: BI 764122 50 mg (Experimental): 5 film-coated tablets of 10 mg BI 764122 (total 50 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
  Interventions: Drug: BI 764122
- SRD part: BI 764122 100 mg (Experimental): 1 film-coated tablet of 100 mg BI 764122 (total: 100 mg) was administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
  Interventions: Drug: BI 764122
- SRD part: BI 764122 200 mg (Experimental): 2 film-coated tablets of 100 mg BI 764122 (total: 200 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
  Interventions: Drug: BI 764122
- SRD part: BI 764122 300 mg (Experimental): 3 film-coated tablets of 100 mg BI 764122 (total: 300 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
  Interventions: Drug: BI 764122
- SRD part: BI 764122 400 mg (Experimental): 4 film-coated tablets of 100 mg BI 764122 (total: 400 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
  Interventions: Drug: BI 764122
- FE part: BI 764122 50 mg fasted/ BI 764122 50 mg fed (Experimental): 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) were administered as single oral dose with 240 mL water after an overnight fast of at least 10 h, followed by wash-out period of at least 7 days followed by 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) administered as single oral dose with 240 mL water after a standardized high-fat, high-calorie breakfast. Food effect (FE) part.
  Interventions: Drug: BI 764122
- FE part: BI 764122 50 mg fed/ BI 764122 50 mg fasted (Experimental): 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) were administered as single oral dose with 240 mL water after a standardized high-fat, high-calorie breakfast, followed by wash-out period of at least 7 days followed by 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) administered as single oral dose with 240 mL water after an overnight fast of at least 10 h. FE part.
  Interventions: Drug: BI 764122
- Placebo (Placebo Comparator): placebo matching in size and weight to corresponding uncoated or film-coated BI 764122 tablets were administered as single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h). Single rising dose (SRD) part.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 764122 — Tablet
  Arms: FE part: BI 764122 50 mg fasted/ BI 764122 50 mg fed; FE part: BI 764122 50 mg fed/ BI 764122 50 mg fasted; SRD part: BI 764122 100 mg; SRD part: BI 764122 12 mg; SRD part: BI 764122 200 mg; SRD part: BI 764122 25 mg; SRD part: BI 764122 300 mg; SRD part: BI 764122 4 mg; SRD part: BI 764122 400 mg; SRD part: BI 764122 50 mg
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 764122 in healthy male subjects following oral administration of single rising doses.

The objective of the food effect (FE) part is to investigate the relative bioavailability of BI 764122 under fed and fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 50 years (inclusive)
* Body Mass Index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Male subjects who meet any of the following criteria from at least 30 days before the first administration of trial medication until 30 days after trial completion:

  * Use of adequate contraception, e.g. use of condom (male subjects) plus any of the following methods (female partners): intrauterine device, hormonal contraception (e.g. implants, injectables, combined oral or vaginal contraceptives) that started at least 2 months prior to first drug administration to the male subject, or barrier method (e.g. diaphragm with spermicide), or surgically sterilised (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy), or postmenopausal, defined as at least 1 year of spontaneous amenorrhea (in questionable cases a blood sample with FSH above 40 U/L and estradiol below 30 ng/L)
  * Sexually abstinent
  * Vasectomised (vasectomy at least 1 year prior to enrolment) in combination with a barrier method (e.g. condom) Unprotected sexual intercourse with a pregnant female partner and sperm donation is not allowed throughout the study and until 30 days after trial completion.

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure (BP), Pulse Rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse as per investigator judgment or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

In addition, the following trial-specific exclusion criteria apply:

- History of acute pancreatitis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder; 2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; 3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization). For more details refer to: http://trials.boehringer-ingelheim.com/

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial investigated safety, tolerability and pharmacokinetics of single rising doses (SRD) of BI 764122 (partially randomized, placebo-controlled, single-blind, parallel (sequential) group design) and its food effect (FE) (randomized, open-label, single-dose, 2-period, 2-sequence crossover design).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria.
  Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 4 mg BI 764122: 4 uncoated tablets of 1 milligram (mg) BI 764122 (total: 4 mg) were administered as single oral dose with 240 milliliter (mL) of water after an overnight fast of at least 10 hours (h). Single rising dose (SRD) part.
- 12 mg BI 764122: 1 film-coated tablet of 10 mg and 2 uncoated tablets of 1 mg BI 764122 (total: 12 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
- 25 mg BI 764122: 2 film-coated tablets of 10 mg and 5 uncoated tablets of 1 mg BI 764122 (total: 25 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
- 50 mg BI 764122: 5 film-coated tablets of 10 mg BI 764122 (total 50 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
- 100 mg BI 764122: 1 film-coated tablet of 100 mg BI 764122 (total: 100 mg) was administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
- 200 mg BI 764122: 2 film-coated tablets of 100 mg BI 764122 (total: 200 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
- 300 mg BI 764122: 3 film-coated tablets of 100 mg BI 764122 (total: 300 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
- 400 mg BI 764122: 4 film-coated tablets of 100 mg BI 764122 (total: 400 mg) were administered as single oral dose with 240 mL of water after an overnight fast of at least 10 h. SRD part.
- BI 764122 50 mg Fasted/ BI 764122 50 mg Fed: 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) were administered as single oral dose with 240 mL water after an overnight fast of at least 10 h, followed by wash-out period of at least 7 days followed by 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) administered as single oral dose with 240 mL water after a standardized high-fat, high-calorie breakfast. Food effect (FE) part.
- BI 764122 50 mg Fed/ BI 764122 50 mg Fasted: 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) were administered as single oral dose with 240 mL water after a standardized high-fat, high-calorie breakfast, followed by wash-out period of at least 7 days followed by 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) administered as single oral dose with 240 mL water after an overnight fast of at least 10 h. FE part.
Period: Treatment Period 1 (SRD and FE Parts)
Arm/Group | Placebo | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | BI 764122 50 mg Fasted/ BI 764122 50 mg Fed | BI 764122 50 mg Fed/ BI 764122 50 mg Fasted
Started | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-out Period (FE Part Only)
Arm/Group | Placebo | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | BI 764122 50 mg Fasted/ BI 764122 50 mg Fed | BI 764122 50 mg Fed/ BI 764122 50 mg Fasted
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (FE Part Only)
Arm/Group | Placebo | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | BI 764122 50 mg Fasted/ BI 764122 50 mg Fed | BI 764122 50 mg Fed/ BI 764122 50 mg Fasted
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were randomized and treated with at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | BI 764122 50 mg Fasted/ BI 764122 50 mg Fed | BI 764122 50 mg Fed/ BI 764122 50 mg Fasted | Total
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 76
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.4 (10.2) | 32.0 (5.8) | 38.7 (8.6) | 32.7 (8.5) | 35.7 (9.3) | 35.7 (5.8) | 31.8 (7.2) | 33.2 (9.8) | 32.8 (9.4) | 40.8 (10.3) | 36.8 (10.3) | 34.3 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 15 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 75
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  White | 16 | 6 | 5 | 5 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 73
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events
Description: Percentage of subjects with drug-related adverse events.
Time Frame: From drug administration until 11 days thereafter for both single rising doses and food effect parts.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Groups:
- 50 mg BI 764122 Fasted: 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) were administered as single oral dose with 240 mL water after an overnight fast of at least 10 hours. Food effect (FE) part.
- 50 mg BI 764122 Fed: 5 film-coated tablets of 10 mg BI 764122 (total: 50 mg) were administered as single oral dose with 240 mL water after a standardized high-fat, high-calorie breakfast. Food effect (FE) part.
Arm/Group | Placebo | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | 50 mg BI 764122 Fasted | 50 mg BI 764122 Fed
Number analyzed (Participants) | 16 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12
Percentage of participants | 6.3 | 0.0 | 16.7 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 8.3 | 8.3

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 764122 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-inf)
Description: Area under the concentration-time curve of BI 764122 in plasma over the time interval from 0 extrapolated to infinity (AUC0-inf).
Time Frame: Within 30 minutes (min) before and 10, 20, 30, 45min and 1 hour (h), 1h 30min, 2, 3, 4, 6, 8, 10, 12, 24, 34, 48, 72, 96 and 120 h post administration.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects from the treated set (TS) who provided data for at least 1 PK endpoint, who were not excluded due to a protocol violation relevant to the evaluation of PK, and who were not excluded due to PK non-evaluability.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol) * hours (h) /Liter (L)
Arm/Group | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | 50 mg BI 764122 Fasted | 50 mg BI 764122 Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12
nanomole (nmol) * hours (h) /Liter (L) | 534 (19.0) | 1530 (33.3) | 2850 (15.1) | 5260 (23.5) | 9810 (14.1) | 19400 (14.4) | 29600 (12.2) | 45700 (17.4) | 6000 (20.5) | 5810 (20.5)

3. Secondary Outcome: Maximum Measured Concentration of BI 764122 in Plasma (Cmax)
Description: Maximum measured concentration of BI 764122 in plasma (Cmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomle (nmol)/ Liter (L)
Arm/Group | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | 50 mg BI 764122 Fasted | 50 mg BI 764122 Fed
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 12
nanomle (nmol)/ Liter (L) | 154 (22.9) | 565 (16.7) | 1280 (35.3) | 2550 (24.9) | 4410 (45.6) | 8090 (19.3) | 13300 (48.4) | 18600 (21.1) | 2610 (46.3) | 1510 (35.3)

ADVERSE EVENTS:
Time Frame: From drug administration until 11 days thereafter for both single rising doses and food effect parts.
Description: Treated set (TS): The treated set included all subjects who were randomized and treated with at least 1 dose of study drug.
Arm/Group | Placebo | 4 mg BI 764122 | 12 mg BI 764122 | 25 mg BI 764122 | 50 mg BI 764122 | 100 mg BI 764122 | 200 mg BI 764122 | 300 mg BI 764122 | 400 mg BI 764122 | 50 mg BI 764122 Fasted | 50 mg BI 764122 Fed
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/16 | 1/6 | 2/6 | 1/6 | 1/6 | 2/6 | 1/6 | 0/6 | 1/6 | 3/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=16) | 4 mg BI 764122 (N=6) | 12 mg BI 764122 (N=6) | 25 mg BI 764122 (N=6) | 50 mg BI 764122 (N=6) | 100 mg BI 764122 (N=6) | 200 mg BI 764122 (N=6) | 300 mg BI 764122 (N=6) | 400 mg BI 764122 (N=6) | 50 mg BI 764122 Fasted (N=12) | 50 mg BI 764122 Fed (N=12)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results.

Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days.

BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT03794323/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT03794323/SAP_001.pdf